CLINICAL TRIAL: NCT02941081
Title: A Novel Nano-iron Supplement (IHAT) to Safely Combat Iron Deficiency and Anaemia (IDA) in Young Children: a Doubleblind Randomised Controlled Trial
Brief Title: A Novel Nano-iron Supplement to Safely Combat Iron Deficiency and Anaemia in Young Children: a Doubleblind Randomised Controlled Trial
Acronym: IHAT-Gut
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: National Nutrition Agency (NaNa), The Gambia (Unknown); Wellcome Trust (Other); King's College London (Other); University of Cambridge (Other); MRC UK Biostatistics Unit (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SCC 1489
Record Dates: First submitted 2016-10-14; First posted 2016-10-21 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Iron Deficiency, Anaemia in Children
Keywords: iron supplement
MeSH Terms: conditions — Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IHAT (Experimental): IHAT arm: novel iron supplement - 1 dose/day single IMP containing IHAT (iron hydroxide adipate tartrate) powder bioequivalent to 12.5 mg elemental iron (i.e. 20 mg Fe taking into account IHAT's relative bioavailability to ferrous sulphate)
  Interventions: Dietary Supplement: IHAT
- ferrous sulphate (Active Comparator): Ferrous sulphate arm: clinical standard of oral iron supplementation - 1 dose/day single IMP containing ferrous sulphate (FeSO4 ) powder equivalent to 12.5 mg elemental iron
  Interventions: Dietary Supplement: Ferrous Sulphate
- placebo (Placebo Comparator): Placebo arm: 'no iron' arm - 1 dose/day containing saccharose powder
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: IHAT — 1 dose/day single IMP containing IHAT powder bioequivalent to 12.5 mg Fe (i.e. 20 mg Fe taking into account IHAT's relative bioavailability to FeSO4)
  Arms: IHAT
Dietary Supplement: Ferrous Sulphate — 1 dose/day single IMP containing FeSO4 powder equivalent to 12.5 mg Fe
  Arms: ferrous sulphate
Other: Placebo — 1 dose/day containing a placebo powder (no-iron, 'sugar' compound)
  Arms: placebo

SUMMARY:
This study aims to determine whether IHAT is non-inferior to ferrous sulphate at correcting iron deficiency and anaemia, and if IHAT does not increase diarrhoea risk in young children living in rural and resource-poor areas of the Gambia.

The study hypothesis is that IHAT will eliminate iron deficiency and improve haemoglobin levels in young children without increasing infectious diarrhoea or promoting inflammation in the gut.

DETAILED DESCRIPTION:
The primary objectives of this trial are: (i) show non-inferiority of IHAT compared to ferrous sulphate for efficacy (in terms of Hb and iron deficiency correction); (ii) show superiority of IHAT compared to ferrous sulphate in terms of moderate-severe diarrhoea (incidence and prevalence); (iii) show non-inferiority of IHAT compared to placebo in terms of prevalence of moderate-severe diarrhoea.

Secondary objectives are: (i) show that IHAT supplementation does not increase enteric pathogen burden; (ii) show that IHAT supplementation is non-detrimental to the gut microbiome; (iii) show that IHAT supplementation does not cause intestinal inflammation; (iv) describe the impact of IHAT supplementation on hospitalisation and morbidity; (v) determine the effect of IHAT supplementation on systemic inflammation; (vi) determine the effect of IHAT supplementation on systemic markers of iron handling.

To investigate the primary and secondary objectives the investigators will conduct a 3-arm, parallel, randomised, double-blind, placebo-controlled, phase 2, clinical trial.

Participants will be iron deficient anaemic young children living in rural communities in the North Bank of the Upper River Division in The Gambia.

The communities and health centres within the study catchment area (Wuli and Sandu districts) will be sensitised to the study. Young children will be identified using the immunisation records at the health centres. At screening, once mothers/guardians of the child have signed the informed consent form, the child will be physically examined by a study nurse and, if the child is considered as generally healthy, their height and weight will be measured and a finger prick blood sample will be collected for Hb and RDT testing. If z-scores are >-3, 7 ≤Hb< 11 g/dL and the RDT is negative, a small venous blood sample will be collected to confirm the Hb levels and determine serum ferritin. A total of 705 eligible children will be randomised into the 3 study arms (n=235 per arm).

In each study arm, the children will be supplemented daily for 12 weeks (84 days) with either placebo, ferrous sulphate or IHAT. Blood and stool samples will be collected at baseline (Day 1) and at day 15 and day 85 during the intervention period. Following the 12 weeks of intervention there will be an additional active follow-up period of 4 weeks without intervention.

Highly trained and experienced field workers will be visiting all children every day during the 12 weeks supplementation period in order to administer the iron supplements or placebo and on these occasions they will check on the children's general health and actively look for signs of malaria and co-infections. If a child shows signs of these infections, the field worker will refer to the study nurse who will perform adequate tests and the child will be offered the appropriate treatment/referral to the next health center. Three times per week, morbidity data (including questions regarding fever, diarrhoea, vomiting, cough, any other illness, appetite and any mediation taken and assessment of body temperature) will be captured. Every week children will be screened using a finger prick blood sample to determine their malaria and Hb status and children found with a positive RDT during the study will be further tested with a blood film and treated according to national guidelines. These visits will continue 4 weeks post intervention to follow-up on AE/SAEs. Any child where Hb falls below 7 g/dL during the follow-up study period will stop the study and will be referred to the next health centre for managemen

ELIGIBILITY:
Inclusion Criteria:

* Age 6-35 mo.
* Free of malaria (RDT negative)
* HAZ, WAZ, WHZ >-3 SD
* IDA defined as 7≤ Hb <11 g/dl AND ferritin<30 μg/L
* Resident in the study area (and planning to remain in the study area for the duration of the trial)
* Ability and willingness to comply with the study protocol (daily intake of supplement and daily study visits with weekly finger prick)
* Informed consent given by parent or guardian

Exclusion Criteria:

* Congenital disorders
* Chronic disease
* Currently participating in another study
* Currently taking iron supplements/multiple micronutrient supplements
* Currently experiencing moderate-severe diarrhoea, defined as those diarrhoea episodes where (i) the child passes more than 5 loose or watery stools per day, (ii) there is blood in the stool (dysentery), or (iii) the child shows signs of clinical dehydration (assessed by the study nurse based on physical signs such as little or no urination, sunken eyes, and skin that lacks its normal elasticity), will usually require treatment (including ORS)

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 645 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
proportion of children with iron deficiency | at 12 weeks
  Proportion of children at 12 weeks with iron deficiency (Cobas analyser). The choice of the marker to use to define iron deficiency will be made at the time of locking the data analysis plan and we will use the most up to date WHO recommendation at the time. But most likely it will be: ferritin <12 mcg/liter, or <30 mcg/liter in the presence of inflammation (CRP>5), and (soluble transferrin receptor - sTfR)/log10 ferritin index >2.
Proportion of children with anaemia | at 12 weeks
  Proportion of children at 12 weeks with anaemia (Medonic analyser). Anaemia is defined as haemoglobin < 11 g/dl.
incidence density' of moderate-severe diarrhea episodes | over 12 weeks
  Incidence density of moderate-severe diarrhoea episodes over the 12 weeks (questionnaire/assessment by study nurse). Incidence density is defined as the number of new episodes of moderate-severe diarrhoea per child over the 12 weeks intervention
period prevalence of moderate-severe diarrhoea | over 12 weeks
  Period prevalence of moderate-severe diarrhea over the 12 weeks (questionnaire/assessment by study nurse). Period prevalence is defined as the proportion of children with at least one episode of moderate-severe diarrhea over the 12 weeks intervention

SECONDARY OUTCOMES:
Alpha diversity and beta diversity of the faecal microbiome | at baseline, 4 weeks and 12 weeks
  Alpha diversity and beta diversity of the faecal microbiome at baseline, 4 weeks and 12 weeks data from MiSeq sequencing of faecal 16S rRNA)
hospitalisation events | over 12 weeks period
  Number of new hospitalization events per child over the 12 weeks (questionnaire
Ratio of enterobacteria/(bifidobacteria+lactobacilli) abundances | at baseline, 4 weeks and 12 weeks
  Ratio of enterobacteria/(bifidobacteria+lactobacilli) abundances in the faecal microbiome at baseline, 4 weeks and 12 weeks (data from MiSeq sequencing of faecal 16S rRNA)
Proportion of children with episodes of respiratory tract infections and malaria | over 12 weeks
  Proportion of children with episodes of respiratory tract infections and malaria over the 12 weeks (questionnaire)
Proportion of children with enteric pathogens | at baseline, 4 weeks and 12 weeks
  Proportion of children with enteric pathogens at baseline, 4 weeks and 12 weeks (targeted qPCR)
Gut inflammation | baseline day 1, day 15 and day 85
  Gut inflammation measured with faecal calprotectin (ELISA)
Longitudinal prevalence of moderate-severe diarrhoea | over 12 weeks
  Longitudinal prevalence of moderate-severe diarrhoea (questionnaire/assessment by study nurse). Longitudinal prevalence is defined as the number of days a child has moderate-severe diarrhea over the 12 weeks intervention
Incidence density of 'bloody' diarrhea per month | per month
  Incidence density of 'bloody' diarrhea per month (questionnaire/assessment by study nurse). Defined as the number of diarrhea episodes with blood in the stool, as a sign of severe intestinal infection, per child-month of observation
Serum C-reactive protein and Alpha-1-acid glycoprotein | baseline day 1, day 15 and day 85
  Serum C-reactive protein and Alpha-1-acid glycoprotein (Cobas analyser). Markers of systemic inflammation
Serum hepcidin | baseline 1day 1, day 15 and day 85
  Serum hepcidin (ELISA). Marker of systemic iron handling
Serum non-transferrin bound iron | baseline day 1, day 15 and day 85
  Serum non-transferrin bound iron (flurescence chemical assay). Marker of systemic iron handling.
Transferrin saturation | baseline5day 1, day 14 and day 85
  Transferrin saturation (Cobas analyser). Marker of systemic iron handling

CONTACTS AND LOCATIONS:
Overall Officials: Dora Pereira, PhD, Principal Investigator — Cambridge University, UK
Locations (1):
- MRC Unit The Gambia, Basse Santa Su, Upper River Division, The Gambia

REFERENCES:
- [Derived] Mohammed NI, Wason J, Mendy T, Nass SA, Ofordile O, Camara F, Baldeh B, Sanyang C, Jallow AT, Hossain I, Faria N, Powell JJ, Prentice AM, Pereira DIA. A novel nano-iron supplement versus standard treatment for iron deficiency anaemia in children 6-35 months (IHAT-GUT trial): a double-blind, randomised, placebo-controlled non-inferiority phase II trial in The Gambia. EClinicalMedicine. 2023 Feb 9;56:101853. doi: 10.1016/j.eclinm.2023.101853. eCollection 2023 Feb. PMID 36880049
- [Derived] de Goffau MC, Jallow AT, Sanyang C, Prentice AM, Meagher N, Price DJ, Revill PA, Parkhill J, Pereira DIA, Wagner J. Gut microbiomes from Gambian infants reveal the development of a non-industrialized Prevotella-based trophic network. Nat Microbiol. 2022 Jan;7(1):132-144. doi: 10.1038/s41564-021-01023-6. Epub 2021 Dec 31. PMID 34972822
- [Derived] Pereira DIA, Mohammed NI, Ofordile O, Camara F, Baldeh B, Mendy T, Sanyang C, Jallow AT, Hossain I, Wason J, Prentice AM. A novel nano-iron supplement to safely combat iron deficiency and anaemia in young children: The IHAT-GUT double-blind, randomised, placebo-controlled trial protocol. Gates Open Res. 2018 Oct 11;2:48. doi: 10.12688/gatesopenres.12866.2. eCollection 2018. PMID 30569038